CLINICAL TRIAL: NCT03168399
Title: A Study to Evaluate the Acceptability of PKU Explore, a Renovated Phenylalanine Free Second Stage Protein Substitute for Use in the Dietary Management of Phenylketonuria in Infants From 6 Months to 5 Years of Age With Regard to Product Tolerance and Adherence.
Brief Title: Evaluation of PKU Explore
Acronym: PKU Explore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Collaborators: Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCT-PKUE-2016-12-05; 219119 (Other: IRAS)
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Phenylketonuria; Inborn Errors of Metabolism
Keywords: Phenylketonuria; PKU; Metabolism; Metabolic; Control; Acceptability
MeSH Terms: conditions — Phenylketonurias; Metabolism, Inborn Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Consumption of PKU Explore (Experimental): Daily feed, substituting the participant's normal phe-free protein substitute for PKU Explore.
  Interventions: Dietary Supplement: PKU Explore

INTERVENTIONS:
Dietary Supplement: PKU Explore — PKU Explore is an unflavoured, powdered, phenylalanine-free, protein substitute, containing essential and non-essential amino acids, carbohydrate, sugar, vitamins, minerals, trace elements and the long chain polyunsaturated fatty acids (LCPs); arachidonic acid (AA) and docosahexaenoic acid (DHA).

SUMMARY:
To evaluate the acceptability, tolerance and effect on metabolic control of PKU Explore, a renovated Phe free protein substitute for the dietary management of PKU in children from 6 months to 5 years.

DETAILED DESCRIPTION:
This is a prospective, acceptability study to evaluate the gastrointestinal tolerance, palatability and adherence of PKU explore in a four-week period for 15 participants aged between 6 months and 5 years for the dietary management of PKU.

The outcome of this assessment will be used in a submission to the regulatory authorities, Advisory Committee on Borderline Substances (ACBS), for PKU Start to become reimbursable on prescription in the UK.

The participant's dietitian will advise on an appropriate amount of PKU Explore based on individual requirements. Parents/carers will be asked to substitute their usual Phe-free protein substitute with PKU Explore for one (1) month. The sponsor will supply PKU Explore free of charge.

Parents/guardians will be asked to record information about the following:

Daily PKU Explore intake Stools Vomiting and Spit-up Feed / Fluid Intake Compliance Phenylalanine Levels (from their routine blood spot testing)

Final Evaluation about the presentation of the product, ease of preparation and use.

ELIGIBILITY:
Inclusion Criteria:

i. A diagnosis of PKU on new-born screening requiring a low protein diet and Phe-free L-amino acid supplements.

ii. Aged between 6 months and 5 years.

iii. Already taking a second stage concentrated protein substitute as part of their PKU management OR is at the stage in their PKU management when a second stage concentrated protein substitute is recommended to commence.

iv. Willingly given, written, informed consent from parent/guardian.

v. Willingly given, written assent (if appropriate).

Exclusion Criteria:

i. Diagnosis of persistent hyperphenylalaninaemia, or mild PKU not requiring dietary treatment with a low protein diet and Phe-free L-amino acid supplements.

ii. Diagnosis of a concurrent condition which may adversely affect developmental progression and feeding ability.

iii. Participation in any other clinical trial/acceptability study.

iv. Any serious medical precluding the study intervention.

v. Use of additional macro/micronutrient supplements during the study period, unless clinically indicated and prescribed by the investigator (must be recorded in patient case record file).

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Product compliance daily diary | Days 1-28
  Quantitative assessments from subject questionnaires that allow evaluation of compliance with the study product, i.e. actual versus prescribed intake.
GI tolerance daily diary assessing change | Days 1-7 and 22-28
  Qualitative assessments from subject questionnaires that allow evaluation of any change in the gastro-intestinal tolerance of the study product.
Ease of use questionnaire | Day 29
  Qualitative assessment from subject questionnaire that allows evaluation of the ease of use of the study product.
Weekly phenylalanine control | Days 1-28
  Collection of quantitative data regarding phenylalanine control using routine biochemical testing

CONTACTS AND LOCATIONS:
Overall Officials: Anita MacDonald, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - NHS Greater Glasgow and Clyde, Glasgow, Lanarkshire
  - Birmingham Women's and Children's NHS Foundation Trust, Burringham, West Midlands
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford, West Yorkshire

IPD SHARING:
Plan to Share IPD: No